CLINICAL TRIAL: NCT02222116
Title: OCT Study of the MGuard Prime Embolic Protection Stent in Patients With Acute ST-segment Elevation Myocardial Infarction
Brief Title: OCT Study of the MGuard Prime Stent in Patients With Heart Attacks
Acronym: MASTER-OCT
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Market move to DES
Sponsor: InspireMD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMD-15
Record Dates: First submitted 2014-08-19; First posted 2014-08-21 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: ST Segment Elevated Myocardial Infarction
Keywords: STEMI; BMS; DES; mesh
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MGuard Prime (Experimental): MGuard Prime
  Interventions: Device: MGuard Prime
- Control (Active Comparator): BMS or DES
  Interventions: Device: Control BMS DES

INTERVENTIONS:
Device: MGuard Prime
  Arms: MGuard Prime
Device: Control BMS DES
  Arms: Control

SUMMARY:
The objective is to demonstrate that the Flow Area within a blocked coronary vessel as assessed by OCT is greater with the MGuard Prime stent compared to non-mesh control stent (BMS/DES) in subjects undergoing primary PCI for ST-segment elevation MI. The study hypothesis is that end of procedure flow area is greater with the MGuard Prime compared with stenting with a non-mesh DES or BMS.

ELIGIBILITY:
Inclusion Criteria:

* Subject is >18 years of age.
* Subject is experiencing clinical symptoms consistent with acute myocardial infarction (AMI) of >30 minutes and ≤12 hours in duration.
* ST-segment elevation ≥1 mm per lead in ≥2 contiguous leads is present in at least one ECG prior to consent.
* Subject agrees to all required follow-up procedures and visits.
* Subject provides written, informed consent.
* The target lesion is a single de novo lesion in a native coronary artery.
* Based on coronary anatomy, PCI is indicated for the culprit lesion with anticipated use of stenting.
* TIMI flow of 0/1 is present at baseline and TIMI flow of 2/3 is present prior to randomization.
* The reference vessel diameter (RVD) of the infarct lesion is 2.75-4.0 mm by visual assessment, assessed after TIMI 2/3 flow is restored.
* The entire lesion length requiring treatment is ≤33 mm by visual assessment, assessed after TIMI 2/3 flow is restored.

Exclusion Criteria:

* Currently enrolled in another investigational device or drug trial that has not reached the primary endpoint or that clinically interferes with the current study endpoints.
* A previous coronary interventional procedure of any kind within 30 days - - - Female patients of childbearing potential.
* Subject undergoing cardiopulmonary resuscitation (patients in whom cardiopulmonary resuscitation was successfully performed and in whom normal mental status was achieved, may be enrolled).
* Cardiogenic shock (SBP <80 mmHg for >30 minutes, or requiring IV pressors or intra-aortic balloon bump (IABP) or other hemodynamic support device for hypotension).
* Prior administration of thrombolytic therapy for the current admission
* Concurrent medical condition with a life expectancy of less than 12 months.
* History of cerebrovascular accident or transient ischemic attack within the last 6 months, or any permanent neurologic deficit
* Prior intracranial bleed at any time, or known intracranial pathology (e.g. tumor, arteriovenous malformation, or aneurysm).
* Active or recent major bleeding within 6 months.
* History of bleeding diathesis or coagulopathy or inability to accept blood transfusions.
* Known hypersensitivity or contraindication to i) aspirin; or ii) heparin and bivalirudin; or iii) clopidogrel, prasugrel and ticagrelor; or iv) cobalt or nickel; or v) contrast media, which cannot be adequately pre-medicated (prior anaphylaxis, however, is an absolute contraindication to enrollment).
* Known calculated creatinine clearance <30 mL/min, hemoglobin <10 g/dL or platelet count <150,000 for the present admission or within 7 days prior to index procedure, if available. NOTE: Baseline labs do not have to be available to consent patient. If laboratory results become available only after randomization, and do not meet inclusion and exclusion criteria, the patient will not be de-registered from the study.
* Surgery planned or any other reason necessitating discontinuation of dual anti-platelet therapy (aspirin and an ADP antagonist) within 6 months.
* Rheolytic thrombectomy, a PTCA balloon with diameter >2.0 mm, or any other device (other than guide wire or simple manual aspiration) is required to restore TIMI 2/3 flow in the infarct vessel.
* Unprotected left main stenosis ≥50% or planned left main intervention.
* Any non-study lesion in the infarct artery with visually estimated diameter stenosis ≥50% and reference vessel diameter ≥2.0 mm or that will require treatment during the index procedure.
* Multi-vessel or multi-lesion intervention required during the index procedure.
* Excessive tortuosity, calcification or diffuse distal disease is present either proximal to, at or distal to the target lesion making it unlikely that the OCT catheter or stent will be able to reach or can be deployed across the target lesion with full expansion.
* Target lesion is a bifurcation with a side branch ≥2.0 mm in diameter.
* Target lesion is at the site of or within a vessel with a previously implanted stent.
* Target lesion is within a bypass graft conduit, or can only be reached by passing the study stent through a bypass graft conduit.
* Aortic dissection or mechanical complication of STEMI (papillary muscle rupture, ventricular septal defect or free wall rupture with or without pseudoaneurysm) identified by left ventriculography or any other modality (such as echocardiography, MRI, CT, physical exam).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10; Primary Completion 2015-11 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is the minFA as measured by OCT at end of primary PCI (after stent deployment but before postdilatation), powered to demonstrate superiority of the MGuard Prime stent compared to the control arm. | immediate

CONTACTS AND LOCATIONS:
Overall Officials: Ori Ben Yehuda, MD, Principal Investigator — CRF; Simon Eccleshall, MD, Principal Investigator — Norfolk and Norwhich Hospitals
Locations (1):
- Norfolk and Norwhich Hospital, Norfolk, United Kingdom